CLINICAL TRIAL: NCT03230110
Title: Obstructive Sleep Apnea Among Pregnant Women With Chronic Hypertension
Brief Title: OSA in Pregnant Women With Chronic HTN
Acronym: OSA-CHTN
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Society for Obstetric Anesthesia and Perinatology (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00081272
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2018-10

CONDITIONS: Sleep Apnea, Obstructive; Pregnancy; Hypertension
Keywords: Sleep disordered breathing; Obstructive sleep apnea; Hypertension; Pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic Hypretension in Pregnancy: Pregnant subjects between 10-20 weeks gestation with chronic hypertension (on medication or hypertensive blood pressures documented at 2 clinic visits)
  Interventions: Diagnostic Test: WP200U home sleep study device
- Normotensive in Pregnancy: Pregnant subjects between 10-20 weeks gestation with normal blood pressure, and not on any treatment for chronic hypertension and no history of chronic hypertension, and matched for body mass index (+/- 3 kg/m2) with the chronic hypertension group.
  Interventions: Diagnostic Test: WP200U home sleep study device

INTERVENTIONS:
Diagnostic Test: WP200U home sleep study device — WP200U, is a Type III, wrist-worn, FDA-approved home sleep testing device that utilizes finger plethysmography (peripheral arterial tone, oxyhemoglobin saturation and heart rate), actigraphy (movement), acoustic decibel detection (snoring volume), and accelerometry (body position) to help diagnose sleep-related breathing disorders (including snoring), and to give information about sleep stages and position during actual sleep time.
  Other Names: WatchPAT

SUMMARY:
The purpose of this study is to identify whether pregnant women with chronic hypertension are at significantly higher risk of having undiagnosed OSA and should be routinely screened with home sleep tests. The investigators will recruit 120 pregnant subjects between 10-20 weeks gestation from the Duke High Risk Obstetrics Clinic over a 20-month period. They will be enrolled into one of two groups: 1) chronic hypertension (on medication or hypertensive blood pressures documented at 3 clinic visits); 2) normal blood pressure, and not on any treatment for chronic HTN and no history of chronic HTN, and matched for BMI (+/- 3 kg/m2) with the chronic HTN group. The two groups will be matched for BMI to control for the effect of obesity on OSA diagnosis and cHTN. The primary hypothesis, that OSA prevalence differs between patients with chronic HTN and normotensive controls, will be assessed with a two-group two-sided Fisher's exact test. A Fisher's exact test with a 0.05 two-sided significance level will have 92% power to detect the difference between a normotensive OSA rate of 0.10 and a chronic hypertensive OSA rate of 0.40 when the sample size in each group is 50. There are no risks associated with the use of the home sleep test device, but subjects that have a severe latex allergy should not participate, as the device

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman who are patients of:Duke Hospital, Duke Birthing Center (DBC), Duke Perinatal Durham clinic, Inpatients will be recruited from the obstetric antepartum service.
* Gestational age 10 weeks, 0 days to 20 weeks, 6 days
* 18 years or older
* English speaking
* They will be enrolled into one of two groups:-Chronic hypertension (on medication or hypertensive blood pressures documented on two clinic visits (including prior to pregnancy), -Normal blood pressure, and not on any treatment for chronic HTN and no history of chronic HTN, and matched for BMI (+/- 3 kg/m2) with the chronic HTN group
* The two groups will be matched for body mass index to control for the effect of obesity on OSA diagnosis and HTN.
* Subjects will be not be excluded if they have an established diagnosis of OSA that is not currently being treated.

Exclusion Criteria:

* Being treated for OSA
* On chronic opioids
* On alpha-blockers (which can interfere with the PAT signal)
* Have secondary HTN
* Unwilling to remove nail polish and/or shorten one nail (which can also interfere with the PAT signal)
* Have a severe allergy to latex
* Do not speak English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Limited to pregnant women
Study Population: The investigators will recruit 120 adult pregnant subjects between 10-20 weeks gestation from Duke Hospital and clinics in Durham, NC over a 20-month period. They will be enrolled into one of two groups: 1) chronic hypertension (on medication or hypertensive blood pressures documented on two clinic visits); 2) normal blood pressure, and not on any treatment for chronic HTN and no history of chronic HTN, and matched for BMI (+/- 3 kg/m2) with the chronic HTN group. The two groups will be matched for BMI to control for the effect of obesity on OSA diagnosis and cHTN.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA in pregnant women with chronic HTN | 20 months
Prevalence of OSA in pregnant women who are normotensive and BMI-matched to women with chronic HTN | 20 months

SECONDARY OUTCOMES:
Apnea-hypopnea indices in pregnant women with untreated OSA and cHTN | 20 months
Apnea-hypopnea indices in pregnant women with untreated OSA and normotensive. | 20 months
Oxygen-desaturation indices in pregnant women with untreated OSA and cHTN | 20 months
Oxygen-desaturation indices in pregnant women with untreated OSA and normotensive. | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dominguez, MD, MHS, Principal Investigator — Duke University Medical Center, Dept Anesthesiology
Locations (2):
- United States (2):
  - Duke Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dominguez JE, Grotegut CA, Wright MC, Habib AS. Obstructive Sleep Apnea Among Gravidas With Chronic Hypertension Compared to Matched Controls: A Prospective Cohort Study. Anesth Analg. 2023 Feb 1;136(2):205-214. doi: 10.1213/ANE.0000000000006223. Epub 2022 Nov 10. PMID 36355613